CLINICAL TRIAL: NCT07251140
Title: Novel Acoustic Biopatch for the Investigation of Dysphagia
Brief Title: Dysphagia Study Using Novel Microphone Device
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Hyojung Choo, Assistant Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00009053; 2025P011062 (Other: Emory IRB)
Record Dates: First submitted 2025-11-03; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Dysphagia; Stroke
MeSH Terms: conditions — Deglutition Disorders; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Novel Acoustic Biopatch for the Investigation of Dysphagia Cohort (Experimental): The device is composed of a sensor (disposable part) and a circuit (reusable part).
  The device will be applied to the anterior neck of dysphagia symptomatic patients who will be accessed with routine dysphagia investigation, such as standard swallowing evaluation with a modified barium swallow (VFSS). Device will be applied by authorized investigators to specific area to target specific neck muscles where no interference occurs for X-ray imaging (VFSS) interpretation. Acoustic data collected via device will be compared with X-ray imaging (VFSS) to train Convolutional neural network (CNN) algorithm to improve accuracy and to determine accuracy of device.
  Interventions: Device: Microphone device

INTERVENTIONS:
Device: Microphone device — * An investigational nanomembrane patch, which is a thin film, is designed to collect acoustics while swallowing.
  * The Microphone is also placed between the thyroid and cricoid cartilages to record swallowing acoustics.

SUMMARY:
This study aims to collect swallowing acoustics with a novel non-invasive wearable surface microphone device during routine work-up, videofluoroscopic swallow study (VFSS), of patients with dysphagia (swallowing trouble). The collected microphone data will be analyzed to find the pattern of abnormal swallowing by machine learning algorithm.

DETAILED DESCRIPTION:
Difficulty swallowing is a very common laryngeal problem affecting many individuals. This study aims to optimize and validate a device to detect dysphagia without invasive procedures. This is an investigational nanomembrane patch, which is a thin film, that will be attached to the subject's chin to check the activity of their muscles. The patch is designed to determine the movement of their muscles and acoustics while swallowing.

This is a prospective cohort study. Dysphagic individuals with stroke visiting Emory University Hospital and Emory Midtown hospital will be asked to participate in the study. Individuals above the age of 40 years will be recruited. The study will be explained in detail to the individuals. After which a written signed consent will be obtained by research personnel before performing any research procedure. The biopatch will be placed and calibrated in dysphagic individuals at the time of performing a barium swallowing test. The collected medical (dysphagia questionnaire) data and demographic data will be collected and saved in Emory REDCap.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis or suspected stroke
* Stroke with additional neurological disorders
* Age between 40 and 85
* Male and Female
* Scheduled to VFSS due to suspected dysphagia, which is determined by bedside water swallowing test and EAT-10 questionnaire as a standard of care.

Exclusion Criteria:

* BMI>35 as an exclusion criteria to recruit participants due to limited transmission of acoustics through increased subcutaneous fat.
* Head and neck cancer treatment history

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10-12 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Normalized Surface Acoustic Swallowing Signal | Up to 30 min post-intervention
  Surface acoustic swallowing signals will be collected using a wearable biopatch containing a microphone, placed on study participants. Raw acoustic data will be recorded in voltage and subsequently normalized against background acoustic levels, resulting in a unitless measure expressed in arbitrary units (a.u.).

SECONDARY OUTCOMES:
Time to apply device to patients | Up to 30 min post-intervention
  Time to apply the device to patients will be recorded in minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Hyojung Choo, PhD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No